CLINICAL TRIAL: NCT07294508
Title: An Open-Label, Randomized, Multicenter, Phase II/III Clinical Study to Evaluate HLX22 (Recombinant Humanized Anti-HER2 Monoclonal Antibody Injection) in Combination With HLX87 (HER2 ADC) as First-Line Treatment in Patients With HER2-Positive Recurrent or Metastatic Breast Cancer
Brief Title: A Study to Evaluate HLX22 in Combination With HLX87 in Patients With HER2-Positive Recurrent or Metastatic Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLX87-BC001
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: HER2 + Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HLX87+ HLX22 (Experimental): Patients will receive the treatment once every 3 weeks (Q3W) until progressive disease (PD) , initiation of new anti-tumor therapy, death, intolerable toxicity, withdrawal of informed consent, or end of the study (whichever occurs first).
  Interventions: Drug: HLX87 + HLX22
- HLX87+ Pertuzumab (Experimental): atients will receive the treatment once every 3 weeks (Q3W) until progressive disease (PD) , initiation of new anti-tumor therapy, death, intolerable toxicity, withdrawal of informed consent, or end of the study (whichever occurs first).
  Interventions: Drug: HLX87 + Pertuzumab
- T-Dxd + Pertuzumab (Active Comparator): Patients will receive the treatment once every 3 weeks (Q3W) until progressive disease (PD) , initiation of new anti-tumor therapy, death, intolerable toxicity, withdrawal of informed consent, or end of the study (whichever occurs first).
  Interventions: Drug: T-Dxd + Pertuzumab
- THP (Active Comparator): Patients will receive the treatment once every 3 weeks (Q3W) until progressive disease (PD) , initiation of new anti-tumor therapy, death, intolerable toxicity, withdrawal of informed consent, or end of the study (whichever occurs first).
  Interventions: Drug: THP

INTERVENTIONS:
Drug: HLX87 + HLX22 — HLX87 is a novel HER2-targeted ADC with a similar mechanism of action to trastuzumab deruxtecan. HLX22 is a novel monoclonal antibody targeting HER2 .
  Arms: HLX87+ HLX22
Drug: HLX87 + Pertuzumab — HLX87 is a novel HER2-targeted ADC with a similar mechanism of action to trastuzumab deruxtecan
  Arms: HLX87+ Pertuzumab
Drug: T-Dxd + Pertuzumab — T-Dxd is a HER2-targeted ADC
  Arms: T-Dxd + Pertuzumab
Drug: THP — Pertuzumab+ Trastuzumab+Docetaxel
  Arms: THP

SUMMARY:
The study is being conducted to evaluate the clinical efficacy of HLX22 in combination with HLX87 as first-line treatment in patients with HER2-positive recurrent or metastatic breast cancer

DETAILED DESCRIPTION:
The study consists of two stages Stage I is an open-label, multicenter, randomized, parallel-controlled phase II clinical study, and its primary objective is to evaluate the clinical efficacy of HLX22 in combination with HLX87 as first-line treatment in patients with HER2-positive recurrent or metastatic breast cancer based on ORR and PFS results.

Stage II is an open-label, multicenter, randomized, parallel-controlled phase III clinical study, and its primary objective is to evaluate the clinical efficacy of HLX22 in combination with HLX87 as first-line treatment in patients with HER2-positive recurrent or metastatic breast cancer based on PFS results.

ELIGIBILITY:
Inclusion Criteria:

* 1. Have a full understanding of the study content, and sign the informed consent form (ICF); 2. Aged ≥ 18 years at the time of signing the ICF, male or female; 3. Histopathologically confirmed breast cancer that meets the following criteria:

  1. Advanced or metastatic breast cancer.
  2. HER2-positive as determined by the central laboratory, defined as IHC 3+, or IHC 2+ and ISH+.
  3. Positive or negative for hormone receptor HR (including estrogen receptor [ER] and progesterone receptor [PgR]) as determined by the central laboratory 4. No prior chemotherapy or HER2-targeted therapy for advanced or metastatic breast cancer (1 line of endocrine therapy is allowed).

  5. At least one measurable lesion as assessed by central imaging according to RECIST v1.1.

  7. Eastern Cooperative Oncology Group performance status score within 7 days prior to the first dose of study drugs: 0-1.

  8. Life expectancy ≥ 12 weeks. 9. Adequate organ functions

Exclusion Criteria:

* 1. History of a second malignancy within 3 years prior to signing the ICF. 2. Previous use of doxorubicin with a concentration of > 360 mg/m2 (or equivalent).

  3. Prior treatment with ADCs including exatecan derivatives that contain topoisomerase I inhibitors.

  4. Uncontrolled or significant cardiovascular diseases 5. Cerebrovascular accidents within 6 months prior to the first dose of study drugs.

  6. ILD/pneumonitis, or suspected ILD/pneumonitis or clinically significant lung-specific intercurrent illness .

  7. Active infection . 8. Presence of spinal cord compression or clinically symptomatic central nervous system metastases.

  9. Residual toxicity from previous anti-tumor therapy that has not resolved to Grade ≤ 1 as per NCI-CTCAE V6.0 or baseline level (except for alopecia).

  10. Presence of active tuberculosis. 11. Have received treatment with live attenuated vaccines within 30 days prior to the first dose of study drugs.

  12. Known history of severe allergic reaction to macromolecular protein preparations, hypersensitivity to the ingredient of the investigational products, or severe hypersensitivity to any excipient of the study drugs.

  13. Known history of abuse of psychotropic drugs or drug addiction. 14. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 706 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2028-01-15 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) (assessed by the blinded independent central review [BICR] as per RECIST v1.1) | up to 26 months
Progression-free survival (PFS) (assessed by BICR as per RECIST v1.1) | up to 37 months

SECONDARY OUTCOMES:
● ORR (assessed by the investigator as per RECIST v1.1) | up to 26 months
● PFS (assessed by the investigator as per RECIST v1.1) | up to 37 months
Second progression-free survival (PFS2) | up to 37 months
Overall survival (OS) | up to 37 months
Incidence and severity of adverse events (AEs) | up to 37 months
  severity determined according to National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version 6.0

CONTACTS AND LOCATIONS:
Overall Officials: Fei Ma, Dr, Principal Investigator — Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China